CLINICAL TRIAL: NCT06109857
Title: Bladder Bank (a Prospective Banking Study)
Status: Recruiting | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Sponsor
Other Study IDs: 21-009854; NCI-2023-00644 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 21-009854 (Other: Mayo Clinic in Rochester)
Record Dates: First submitted 2023-10-25; First posted 2023-10-31 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Bladder Carcinoma
MeSH Terms: conditions — Urinary Bladder Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood Collection: At study enrollment for subjects, 60 ml (4 tablespoons) of blood will be drawn from all participants and will be processed according to standardized study biospecimen protocol. Specimens will be stored in a secure lab for future approved research.
  Urine Collection: At study enrollment for subjects, up to 20mL of urine in 5 ml aliquots (stored with or without fixative in up to 5 equal aliquots) from the same or unique case patients above targeted for blood collection.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Observational: Patients undergo blood and urine sample collection and have their medical records reviewed while on study.
  Interventions: Other: Non-Interventional Study

INTERVENTIONS:
Other: Non-Interventional Study — Non-interventional study

SUMMARY:
This study collects blood and urine samples from patients with bladder cancer to support the development of tests for early detection of bladder cancer.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To establish a biobank of samples (blood and urine) to support the development of non-invasive tests for early detection of bladder cancer.

OUTLINE: This is an observational study.

Patients undergo blood and urine sample collection and have their medical records reviewed while on study.

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years
* Patient has undergone office-based evaluation for hematuria [computed tomography (CT), ultrasound, cystoscopy]

Exclusion Criteria:

* Patient has known cancer outside of the target cancer 5 years prior to current collection (not including basal cell or squamous cell skin cancers; if patient has not been seen or if information is not available, the patient is eligible)
* Patient has recurrent muscle invasive bladder cancer
* Patient has ever been previously diagnosed with UTUC (upper tract urothelial carcinoma) prior to bladder resection
* Patient has received chemotherapy class drugs for the treatment of non-target origin cancer in the 5 years prior to current collection
* Patient has had any prior radiation therapy to the target lesion prior to current collection
* Patient has had a biopsy to the target organ and/or lesion within 3 days before collection
* Patient has undergone cystectomy or cystoprostatectomy
* Patient has transurethral instrumentation (placement of urinary catheter) within 7 days prior to urine collection
* Patient has had a urinary tract infection within 14 days prior to urine collection
* Patient has chronic indwelling urinary catheter

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient has undergone office-based evaluation for hematuria
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2022-07-06 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Blood sample to support the development of non-invasive tests for early detection of bladder cancer | Baseline (at enrollment)
  At study enrollment for subjects, 60 ml (4 tablespoons) of blood will be drawn from all participants and processed according to standardized study biospecimen protocol. All samples will be stored for future analysis in Molecular Cancer Diagnostic Laboratory at Mayo Clinic.
Urine sample to support the development of non-invasive tests for early detection of bladder cancer | Baseline (at enrollment)
  At study enrollment for subjects, up to 20mL of urine will be collected from the same or unique case patients identified for blood collection. All samples will be stored for future analysis in Molecular Cancer Diagnostic Laboratory at Mayo Clinic.

CONTACTS AND LOCATIONS:
Overall Officials: John B. Kisiel, MD, Principal Investigator — Mayo Clinic in Rochester
Locations (1):
- Mayo Clinic in Rochester, Rochester, Minnesota, United States

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials